CLINICAL TRIAL: NCT01719965
Title: Evaluation of the Tak Province Community Ethics Community Advisory Board: Interviews and Focus Group Discussions
Brief Title: Evaluation of Tak Community Advisory Board
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: CTSG1201
Record Dates: First submitted 2012-10-17; First posted 2012-11-01 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Community Members
Keywords: Community Advisory Board; Focus Group Discussion; Interview; Community Engagement; Thailand
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Health Workers: * Worked in SMRU for at least 6 months
  * Clinic assistants, medics or home visitors
  Interventions: Other: Interviews and Focus Group Discussions
- Researchers: * Worked in SMRU for at least 6 months
  * Physician or scientist
  Interventions: Other: Interviews and Focus Group Discussions
- CAB members: - Member of the CAB for at least 3 months
  Interventions: Other: Interviews and Focus Group Discussions
- Community members: - Lived in the border area (area served by SMRU or Mae Sot) for at least 6 months
  Interventions: Other: Interviews and Focus Group Discussions
- Research subjects: - Participants who are currently enrolled in an SMRU study
  Interventions: Other: Interviews and Focus Group Discussions

INTERVENTIONS:
Other: Interviews and Focus Group Discussions

SUMMARY:
A popular form of community engagement is for the researchers to interact with a Community Advisory Board. The Shoklo Malaria Research Unit has been working on the Thai-Burmese border for many years and has been informally engaging with the community for its healthcare and research initiatives, especially in the area of ethics and consent. In January 2009, community engagement was formalised with the establishment of the Tak Province Border Community Ethics Advisory Board (T-CAB). The T-CAB is the first of its kind as the investigators have not come across any set up of similar nature involving mobile and unstable populations residing along a porous border.

Three years on, SMRU questions if the T-CAB has been "successful" and if the current T-CAB model is the best model for this community. In order to evaluate the T-CAB, first an evaluation tool has to be developed as there are no off-the-shelf evaluation tools for CABs, then the evaluation will be carried out.

DETAILED DESCRIPTION:
1. Background

Research on the Thai-Myanmar border

Since 1986, the Shoklo Malaria Research Unit (SMRU) has provided basic healthcare and carried out research aimed at reducing the impact of multi-drug resistant malaria and other infectious diseases in the area on the border between Thailand and Myanmar. SMRU's main area of interest is in malaria, with special interest in children and pregnant women - the groups most at risk from malaria - and it has combined this research with the operation of antenatal clinics along the border. SMRU currently runs multiple free clinics for the Karen and Burman border population that would otherwise lack access to health care. The most distant clinic is about 120 km from the SMRU office in Mae Sot. Carrying out research and providing care along the border presents a range of unique practical and ethical challenges. This in part because the people who live near the border are mostly migrants or refugees from elsewhere in Myanmar who have, since the 1980s, moved to the border area to escape economic hardship and sometimes conflict and persecution. There are currently thought to be two million migrants from Myanmar living in Thailand (about 150 000 in refugee camps) and a further million 'internally displaced' people living near the border inside Myanmar, although numbers are difficult to verify. The vast majority of these people, who come from a very diverse range of different ethnic, religious, political and language groups, live in insecure, unsafe conditions and face a number of serious health difficulties.

Until 1995, SMRU focused its activities primarily in the refugee camps in the border area and a strong collaboration was established with non-govermental organisations (NGOs) to control malaria in the refugee population through the operation of "the Malaria Task Force" (MTF). This was largely successful and malaria is now a minor problem within the camps. As a consequence, whilst SMRU remains responsible for antenatal and obstetric care and the treatment of malaria patients in refugee camps such as Mae La, since 1995 it has increasingly extended its activities to reach out to the wider displaced populations who have little alternative access to malaria diagnosis and treatment or antenatal care. This is done in collaboration with the Thai Ministry of Public Health (MOPH) and in close collaboration with the district hospitals and the Tak provincial health authorities. In 2001-2003 the Tak Malaria Initiative, supported by the Bill & Melinda Gates Foundation deployed the malaria control strategy developed by SMRU in the refugee camps to all 200 affected villages in the province's border districts with substantial success. When the funding from the Gates Foundation came to an end, the MOPH took over the program.

The border between Thailand and Myanmar is at the forefront of the global fight against malaria because it is on the frontline in the battle against the development and spread of resistance to anti-malarial drugs. Malaria parasites found here are some of the most drug-resistant on earth and their expansion and spread is a very real global threat (research has already demonstrated that the most drug-resistant malaria parasites found in Africa originated in South East Asia) . This is particularly urgent and important in the populations living along the border because there is published evidence that the malaria parasites may become tolerant even to the most advanced artemisinin combination therapies (ACTs) now at the forefront of global malaria treatment.

Rationale for the establishment of the community advisory board

There is widespread agreement on the need for community engagement in clinical research, particularly where the research involves minority groups and other vulnerable populations. However there has been little research on the effectiveness and challenges associated with different forms of engagement, and little or no evidence base on which to base engagement strategies.

A popular form of community engagement is for the researchers to interact with a Community Advisory Board. The Shoklo Malaria Research Unit has been working on the Thai-Burmese border for many years and has been informally engaging with the community for its healthcare and research initiatives, especially in the area of ethics and consent. In January 2009, community engagement was formalised with the establishment of the Tak Province Border Community Ethics Advisory Board (T-CAB). The T-CAB is the first of its kind as the investigators have not come across any set up of similar nature involving mobile and unstable populations residing along a porous border.

At the time of its establishment, the T-CAB had three main goals. The first of these was that, after a period of training - about diseases such as malaria and the nature and goals of research - it's members would be able to advise on whether a study is acceptable to and perceived as beneficial by, the communities in the region. The second was that, the T-CAB would play a key role in advising researchers on the ethical and operational aspects of proposed studies such as: informed consent procedures, fair compensation, risks and benefits, how to protect the confidentiality of research subjects, and so on. The third, aim was that the T-CAB would act as a 'bridge' between the communities and researchers. It would on the one hand, provide communities with an opportunity to express views on proposed research and to influence and direct research aims, and on the other, provide a means by which the researchers might feedback the results of the research to the community.

Three years on, SMRU questions if the T-CAB has been "successful" and if the current T-CAB model is the best model for this community. In order to evaluate the T-CAB, first an evaluation tool has to be developed as there are no off-the-shelf evaluation tools for CABs, then the evaluation will be carried out.

ELIGIBILITY:
Inclusion Criteria:

A. Health workers

* Worked in SMRU for at least 6 months
* Clinic assistants, medics or home visitors

B. Researchers

* Worked in SMRU for at least 6 months
* Physician or scientist

C. CAB members

- Member of the CAB for at least 3 months

D. Community members - Lived in the border area (area served by SMRU or Mae Sot) for at least 6 months

E. Research subjects

- Participants who are currently enrolled in an SMRU study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community members who work in Tak Province, Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Qualitative Assessment of Community Advisory Board. A summary of opinions raised in interviews. | 90 Minutes
  Individual interviews and Focus Group Discussions. This is an observational study and the outcomes will be the comments the investigators receive from participants. The investigators will bring these views together and highlight general views and any particular points of note or problems identified by participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand